## The First Affiliated Hospital of Shandong First Medical University (Shandong Provincial

## Qianfoshan Hospital)

## Medical Ethics Committee Approval Reports

Lot No.: YXLL-KY-2023(018)

Date: February 25, 2023

| Applicant/Development Unit: The First Affiliated Hospital of Shandong First Medical University | | | | | |
|---|---|---|---|---|---|
| (Shandong Provincial Qianfoshan Hospital) | | | | | |
| Clinical Research Program Number: V2.0 | | | Drug registration lot number: | | |
| Clinical Research Leader: Yan Li | | | | | |
| Clinical Study Title: Effect of Azole/Echinocandin Use on Tacrolimus Pharmacokinetics in Kidney | | | | | |
| Transplant Patients | | | | | |
| Clinical Research Unit and Address: The First Affiliated Hospital of Shandong First Medical University | | | | | |
| (Shandong Provincial Qianfoshan Hospital), No. 16766, Jingshi Road, | | | | | |
| Jinan, China | | | | | |
| Name and Address of the Ethics Committee: Medical Ethics Committee of the First Affiliated Hospital of | | | | | |
| Shandong First Medical University (Shandong Provincial | | | | | |
| Qianfoshan Hospital), No. 16766, Jingshi Road, Jinan, China | | | | | |
| Submissio | Drug Registration Approval | No | Content | Applicant's Qualification | meet the |
| -n of | | | of the | Certificate | requirements |
| materials | Clinical Research Program | Yes | review | Methods of Obtaining | proper |
| | | | | Informed Consent | |
| | Researcher's Handbook | No | | Opinion on the Research | acceptance |
| | | | | Program | |
| | Patient Informed Consent | No | | Review Pathway | Expedited review |
| | Drug Test Compliance Report | No | | | |
| | Case Report Form | Yes | | | |
| | Attachment | Yes | | | |
| Conclusion | Consent | • | | | |
| Ethics Committee Approval Opinion | | | | | |

Ethics Committee Approval Opinion:

The lead reviewer of the ethics committee reviewed and discussed the project in strict accordance with GCP principles and relevant Chinese regulations and guidelines. Based on the results of the review, this committee agreed to carry out the research of this project from the date of approval, and requested the investigator and the sponsor to strictly abide by the National CFDA "Good Clinical Practice (GCP) for Drug Clinical Trials", conscientiously accept the constraints of the relevant national laws and regulations, and pay attention to the prevention of adverse effects and the protection of patients' rights and interests and safety. All information shall not be modified without the approval of the Committee; if any serious adverse events occur in the study, please notify the Committee immediately.

Signature of the Director of the Ethics Committee:



Seal of the Ethics Committee: